CLINICAL TRIAL: NCT02454335
Title: Comparison of Outcome and Complications of Anterior Versus Posterior Myotomy in Per-oral Endoscopic Myotomy (POEM) Endoscopic Procedure for Treatment of Achalasia: Randomized Single Blinded Clinical Trial
Brief Title: POEM Anterior Versus Posterior Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00093759
Record Dates: First submitted 2015-05-10; First posted 2015-05-27 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior Approach (Active Comparator): For the anterior approach, an incision will be made in the 1 to 2 o'clock position of the esophageal wall.
  Interventions: Procedure: Peroral Endoscopic Myotomy
- Posterior Approach (Active Comparator): For the posterior approach, a mucosal incision will be made at the 5 to 6 o'clock position
  Interventions: Procedure: Peroral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Peroral Endoscopic Myotomy — The intervention is the POEM procedure performed by either anterior approach or posterior approach orientation of the incision for mucosal entry.
  Other Names: POEM

SUMMARY:
Per-oral endoscopic myotomy (POEM) is an incisionless procedure used to treat esophageal achalasia, performed by GI endoscopist without cutting any surface of the human body. The main constituent of the procedure is the myotomy part, through which the endoscopist cuts the muscle fibers in the submucosa. Since this procedure is completely new to the area of treatment of achalasia, it is unknown whether a posterior or an anterior myotomy is better in relieving the symptoms. Thenceforth, this study aims at randomizing patients with achalasia presenting for POEM to getting either the posterior or the anterior myotomy. Patients will be followed up for symptoms and complications; data will be extracted and the appropriate analysis will be employed to determine if there is any difference of outcome between the two techniques of myotomy.

DETAILED DESCRIPTION:
Peroral Endoscopic Myotomy (POEM) is an effective, minimally-invasive treatment for achalasia that has been adopted over the past few years. As more programs attempt to adopt the novel technique, there is an increased need for trials to help guide the growth of the procedure. Review of the current literature reveals that most endoscopists prefer an anterior approach, with an incision in the anterior/ anterolateral wall of the esophagus. This approach has been used with tremendous success in decreasing the symptoms of dysphagia and lowering esophageal sphincter (LES) pressure since the first description of the procedure in humans in 2010. However, it can be technically challenging in patients with anterior scarring from prior surgery or radiation, in whom a posterior approach has typically been used. Alternatively, the posterior approach, with incision in the posterolateral wall of the esophagus, has been adopted with great success by several endoscopists as the primary approach to myotomy. Reports involving the posterior approach have also shown significant symptom relief as defined by symptoms score (Eckardt score) < 3, decreased LES pressure, and low complication rates.

However, despite high rates of technical and clinical success, the posterior approach has not been as widely adopted as the anterior approach. Without comparison of the two approaches in terms of efficacy and safety, the optimal technique to myotomy for POEM is yet to be defined. The investigators main hypothesis is that the posterior myotomy is as efficacious as the anterior myotomy in terms of improvement of achalasia symptoms as indicated by reduction in the Eckardt score and LES pressure. Adaptation of both techniques may increase options in approach for routine POEM and increase the number of patients that are able to undergo the procedure, thereby promoting its applicability.

ELIGIBILITY:
Inclusion Criteria for Participants

* Adult patient age greater than 18 years old
* Confirmed diagnosis of achalasia via high resolution esophageal manometry (HREM)

Exclusion Criteria

* Previous surgery of the esophagus or stomach
* Active severe esophagitis
* Large lower esophageal diverticula
* Large > 3cm hiatal hernia
* Sigmoid esophagus
* Known gastroesophageal malignancy
* Inability to tolerate sedated upper endoscopy due to cardiopulmonary instability, severe pulmonary disease or other contraindication to endoscopy
* Cirrhosis with portal hypertension, varices, and/or ascites
* Pregnant or breastfeeding women (all women of child-bearing age will undergo urine pregnancy testing)
* Acute gastrointestinal bleeding
* Uncorrectable coagulopathy defined by INR > 1.5 or platelet < 50

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Eckardt Score | up to 24 months
  The standardized clinical scoring system for achalasia will be assessed at 2 weeks, 3 months, 6 months, and 1 year post procedure. The score is based on the results of a self- administered questionnaire using 4 items related to digestive symptoms including weight loss, dysphagia, retrosternal pain, and regurgitation. Each item is rated from 0 to 3 (0= none, 1= occasional, 2=daily, 3=with every meal).

SECONDARY OUTCOMES:
Rate of GERD by pH-impedance | up to 24 months
  This is assessed by the DeMeester score. The score is comprised of the following: Percent total time pH < 4, Percent Upright time pH < 4, Percent Supine time pH < 4, Number of reflux episodes, Number of reflux episodes ≥ 5 min, Longest reflux episode (minutes). The abnormal reflux is defined as DeMeester score >14.72
Quality of Life by QoL S36 questionnaire | up to 2 years
  The SF-36 general health questionnaire consists of 36 questions evaluating the patient's perception of their quality of life (QoL) in the following eight subscales: physical functioning (PF), role limitations due to physical problems (RP), role limitations due to emotional problems (RE), energy/fatigue (EF), emotional well-being (EW), social functioning (SF), bodily pain (BP) and general health (GH). Subscale scores range from 0 to 100, with 100 being the best and 0 being the worst quality of life.
Dysphagia by the Dysphagia Score | up to 24 months
  Dysphagia scoring system scores dysphagia as follows:
  0 = able to eat normal diet / no dysphagia; 1 = able to swallow some solid foods; 2 = able to swallow only semi solid foods; 3 = able to swallow liquids only; 4 = unable to swallow anything / total dysphagia.
Postoperative pain by VAS analogue scale | 2 years
  The visual analogue scales scores the severity of the pain from zero (minimum) to 10 (maximum).
Analgesic use by Analgesic Quantification Algorithm | up to 24 months
  Analgesic Quantification Algorithm scoring scores analgesic use from zero (minimum) to 7 (maximum) as follows:
  0= No analgesic; 1= Non-opioid analgesics; 2= Weak opioids (For example, codeine and tramadol); 3= Strong opioids ≤75 mg OME per day; 4= Strong opioids >75-150 mg OME per day; 5= Strong opioids >150-300 mg OME per day; 6= Strong opioids >300-600 mg OME per day ; 7=Strong opioids >600 mg OME per day
Operative and post-operative complications | up to 2 years
Hospital stay in days | up to 24 months
LES pressure by Manometry | up to 2 years
Total procedure time and times of different steps | up to 24 months
Technical success | up to 24 months
  Defined as completion of the procedure using the assigned approach
Ease of procedure measured by the Lickerdt scale | up to 24 months
  The ease of the procedure scored by the endoscopist on a Likert scale rated from 1 (easy) to 5 (impossible).

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Khashab MA, Sanaei O, Rivory J, Eleftheriadis N, Chiu PWY, Shiwaku H, Ogihara K, Ismail A, Abusamaan MS, El Zein MH, Wong VW, Billioux VG, Kumbhari V, Kalloo AN, Ponchon T, Pioche M. Peroral endoscopic myotomy: anterior versus posterior approach: a randomized single-blinded clinical trial. Gastrointest Endosc. 2020 Feb;91(2):288-297.e7. doi: 10.1016/j.gie.2019.07.034. Epub 2019 Aug 10. PMID 31408652